CLINICAL TRIAL: NCT01197872
Title: Phase II: Clinical Use of Parental Support To Detect Single Gene Mutations
Brief Title: Clinical Use of Parental Support To Detect Single Gene Mutations
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Matthew Rabinowitz, PhD/ CEO and President, Gene Security Network
Other Study IDs: IVF008.5
Record Dates: First submitted 2010-09-03; First posted 2010-09-09 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Single Gene Disorders
MeSH Terms: interventions — Prostaglandins D; Fertilization in Vitro

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, cheek swab/saliva samples, sperm samples, embryo biopsy samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Preimplantation Genetic Diagnosis — Genetic testing on embryos to identify embryos that are affected by a single gene disorder (e.g. cystic fibrosis, Tay-Sachs, sickle cell anemia).
  Other Names: PGD; In Vitro Fertilization; IVF; Parental Support; Gene Security Network

SUMMARY:
Gene Security Network has developed a novel technology called Parental Support (PS) which is used for Preimplantation Genetic Screening/Diagnosis (PGS/D) during in vitro fertilization (IVF). This technology allows IVF physicians to identify embryos, prior to transfer to the uterus, which have the best chance of developing into healthy children.

DETAILED DESCRIPTION:
This study follows previous IRB approved study IVF008: Clinical Use of Parental Support To Detect Single Gene Mutations , which we will refer to as "Phase I".

The purpose of Phase I was to validate clinical use of PS to detect specific genetic mutation(s) known to cause severe inheritable diseases in embryos produced by at-risk couples, while simultaneously testing these embryos for aneuploidy. The Phase I study consisted of first of its kind PGS/D testing to detect disease-associated genetic mutations together with aneuploidy screening.

This study, which we will call "Phase II", will allow patients to continue to access testing while clinical data is collected on Phase I. Phase I of the study is nearing enrollment targets (40+ participating couples) and Phase I enrollment will be closed while subjects complete testing and study data is collected from pregnancies and livebirths. Phase II will allow: 1) additional data collection prior to commercial testing launch, 2) eligible patients to participate and receive testing.

ELIGIBILITY:
Inclusion Criteria:

At risk couple (mother and father) who are:

* Able to provide laboratory report from commercial CLIA certified laboratory in the United States or legitimate non-US laboratory confirming presence of disease associated mutation in mother and/or father
* Planning to go through IVF and desiring PGD for the specified mutation
* Planning to pursue Chorionic Villus Sampling (CVS) or Amniocentesis if pregnancy occurs and willing/able to provide CVS/ Amniocentesis sample to GSN for confirmatory testing or provide test results of confirmatory testing performed by an external laboratory.

Exclusion Criteria:

* Couples without prior documentation of genetic mutation as specified above
* Couples where the male partner is not willing, able, or available to provide a semen sample
* Unwilling to have CVS/ Amniocentesis
* In certain cases, unavailability of child sample or other suitable family member: Subjects will not be able to enroll in the study if, in the judgment of the research staff, validation is first required on a child (offspring of male and female subject) and there is no child or other family member that is a suitable substitute available for testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Couples in which both parents are carriers or one parent is affected by an inherited condition that they are at risk of passing on to their offspring. These couples must be planning to use In Vitro Fertilization (IVF) and Preimplantation Genetic Diagnosis (PGD).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Confirmation of diagnosis through prenatal diagnosis | 10-20 weeks post intervention
  Confirmation of PGS test results through prenatal diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rabinowitz, PhD, Principal Investigator — CEO, Gene Security Network
Locations (1):
- Gene Security Network, Redwood City, California, United States